CLINICAL TRIAL: NCT03576690
Title: Expanded Access Protocol for Emergency Use of REGN3470-3471-3479 for the Treatment of Ebola Virus Disease
Brief Title: R3470-3471-3479 (REGN-EB3) Expanded Access Protocol (EAP) for Treatment of Ebola Virus Disease
Status: Available | Type: Expanded Access
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: R3470-3471-3479-EBOV-1846
Record Dates: First submitted 2018-06-22; First posted 2018-07-03 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Ebola Virus Disease
Keywords: Positive Ebola Virus (EBOV) diagnostic test; symptomatic
MeSH Terms: conditions — Hemorrhagic Fever, Ebola | interventions — atoltivimab, maftivimab, and odesivimab-ebgn drug combination

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Biological: REGN3470-3471-3479
  Other Names: REGN-EB3; Inmazeb®; atoltivimab, maftivimab, and odesivimab

SUMMARY:
Provide access to REGN-EB3 for the treatment of patients with Ebola Virus Disease (EVD).

ELIGIBILITY:
Key Inclusion Criteria:

* Males or females in an Ebola endemic region with documented positive polymerase chain reaction (PCR) for Ebola virus infection who are symptomatic
* Ability to provide informed consent personally or by a legal representative if the patient is unable to do so, based on local laws and regulations
* REGN-EB3 can be administered to pregnant women infected with Zaire ebolavirus, as defined in the protocol
* Children of any age will be eligible for enrollment, as defined in the protocol
* Neonates born to an infected mother who has not yet cleared the Ebola virus are eligible for enrollment, as defined in the protocol

Key Exclusion Criteria:

* Negative EBOV diagnostic test result
* A patient who, in the judgment of the investigator, will be unlikely to comply with the requirements of this protocol
* Any serious medical condition that, in the opinion of the site investigator, would place the patient at an unreasonable increased risk through participation in this study, including any past or concurrent conditions
* Eligible for an ongoing randomized clinical trial with REGN-EB3

NOTE: Other protocol defined inclusion / exclusion criteria apply

Sex: All
Age Groups: Child, Adult, Older Adult